CLINICAL TRIAL: NCT00036491
Title: An Open-Label Safety and Efficacy Study of an Anti-CD20 Antibody (Rituximab, Rituxan®) for Anti-B Cell Therapy in the Treatment of Systemic Lupus Erythematosus
Brief Title: Anti-CD20 in Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Autoimmunity Centers of Excellence (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT AC002; SACCC #ASL02 (Other: Statistical and Clinical Coordinating Center); UPenn #U1131s (Other: University of Pennsylvania); ACE Study #AC002 (Other: Autoimmunity Centers of Excellence)
Record Dates: First submitted 2002-05-10; First posted 2002-05-13 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Lupus Erythematosus, Systemic
Keywords: Systemic Lupus Erythematosus; SLE; B-Lymphocytes; anti-CD20; rituximab
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- rituximab (Experimental): 375 mg/m^2 administered intravenously
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — Subjects received four weekly infusions of rituximab at a dose of 375 mg/m^2
  Other Names: Rituxan®

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of rituximab (anti-CD20) in treating systemic lupus erythematosus (SLE).

White blood cells in the body called B cells give off substances that are active in promoting SLE disease. Researchers have found that anti-CD20 can block production of these substances in another disease. This study explores whether anti-CD20 will also be safe in people with SLE and whether it may be effective in treating SLE.

DETAILED DESCRIPTION:
B cells clearly play an essential role in the pathogenesis of SLE since they produce autoantibodies. Clinical observations support the contention that intervening in the production of autoantibodies by the B lymphocyte will be effective therapy. Current approved therapy for B-cell non-Hodgkin's lymphoma includes anti-CD20. The results of anti-CD20 administration in SLE are anticipated to be similar to those in lymphoma patients. The current proposal explores the mechanisms and applicability of B-cell depletion as a potential treatment for SLE.

Participants receive 4 weekly infusions of study medication. Each participant is enrolled in the study for a total of 1 year with protocol visits weekly for the first 3 months, then every other week for the next 2 months, every month for the next 4 months, and every other month for the remaining 5 months of the study (Weeks 0, 1, 2, 3, 4, 5, 6, 7, 9, 11, 13, 15, 19, 23, 27, 31, 39, 47, and 55). Responses to exogenous antigens are measured; assessments for clinical response with SLE-disease activity score (SLEDEI) and systemic lupus activity measure (SLAM) score are performed. Participants complete a health questionnaire and a health survey and laboratory parameters are evaluated.

ELIGIBILITY:
Inclusion Criteria

People may be eligible for this study if they:

* Are 18 to 70 years of age
* Agree to use a reliable method of birth control during treatment and for 6 months after treatment ends
* Have SLE (by the American College of Rheumatology criteria)
* Have had SLE for at least 6 months prior to screening
* Have active SLE disease at the screening visit
* Have organ disease (lung, stomach, intestinal, blood, kidney, and/or heart)
* Have failed standard therapy, including at least 1 immunosuppressive agent, or have experienced side effects from an immunosuppressive agent that required discontinuation of treatment
* Meet blood, liver, and kidney laboratory values set by the protocol
* Have not taken an immunosuppressive agent for 2 weeks prior to the first treatment
* Have been on a stable dose of oral corticosteroids, if taking them, for 4 weeks before the first week's visit. Oral corticosteroids may be altered as medically necessary after enrollment.
* Have at least 1 elevated autoantibody level at screening visit.

Exclusion Criteria

People will not be eligible for this study if they:

* Are pregnant or breast-feeding
* Have heart, lung, nervous system, kidney, liver, stomach, intestinal, or other diseases that may place the patient at risk if participating in the trial
* Have cranial neuropathy (a condition affecting the head region)
* Are on blood-thinning agents to prevent blood clotting
* Have a serious skin disease
* Have a certain class of heart disease
* Have had cancer, unless surgically cured basal cell carcinoma or cervical dysplasia
* Have a long term serious infectious disease such as tuberculosis or a fungal infection that is now active, or active within 2 years of the baseline visit
* Have had HIV infection or another immunosuppressive state (chemotherapy or radiation therapy)
* Have received any experimental drug within 30 days of baseline visit
* Have received any monoclonal antibody or similar medication within 3 months of the baseline visit
* Received any intravenous, joint, or muscle injection of corticosteroids within 4 weeks of the baseline visit
* Abuse alcohol or drugs
* Are unwilling or unable to follow the protocol
* Have poor veins for receiving injections.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2001-01; Primary Completion 2006-01 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Serum Autoantibodies | Baseline, Week 4, Week 12, Week 24, Week 36 and Week 56
Systemic Lupus Erythematosus Disease Activity Index (SLEDAI) | Baseline, Week 4, Week 7, Week 11, Week 15, Week 19, Week 27, Week 39 and Week 55

SECONDARY OUTCOMES:
C3 and C4 complement levels
Systemic Lupus Activity Measure (SLAM) | Baseline, Week 4, Week 7, Week 11, Week 15, Week 19, Week 27, Week 39 and Week 55
Erythrocyte Sedimentation Rate (ESR)
Prednisone Dose | Baseline, Week 4, Week 12, Week 24, Week 36 and Week 56
Renal Function
  Measured by creatinine clearance and total protein.
Modified Health Assessment Questionnaire (HAQ)
Short Form-36 Health Survey (SF-36)
Physician Global Assessment (VAS)
Patient Global Assessment (VAS)
Systemic Lupus Erythematosus International Collaborating Clinics (SLICC)/American College of Rheumatology (ACR) Damage Index for SLE
Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Eisenberg, MD, Study Chair — University of Pennsylvania
Locations (3):
- United States (3):
  - University of Colorado, Denver, Colorado
  - University of Rochester, Rochester, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Eisenberg R. Targeting B cells in SLE: the experience with rituximab treatment (anti-CD20). Endocr Metab Immune Disord Drug Targets. 2006 Dec;6(4):345-50. doi: 10.2174/187153006779025757. PMID 17214580
- [Background] Sutter JA, Kwan-Morley J, Dunham J, Du YZ, Kamoun M, Albert D, Eisenberg RA, Luning Prak ET. A longitudinal analysis of SLE patients treated with rituximab (anti-CD20): factors associated with B lymphocyte recovery. Clin Immunol. 2008 Mar;126(3):282-90. doi: 10.1016/j.clim.2007.11.012. Epub 2008 Jan 15. PMID 18226586
- [Result] Albert D, Dunham J, Khan S, Stansberry J, Kolasinski S, Tsai D, Pullman-Mooar S, Barnack F, Striebich C, Looney RJ, Prak ET, Kimberly R, Zhang Y, Eisenberg R. Variability in the biological response to anti-CD20 B cell depletion in systemic lupus erythaematosus. Ann Rheum Dis. 2008 Dec;67(12):1724-31. doi: 10.1136/ard.2007.083162. Epub 2008 Feb 4. PMID 18250115
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov
- Available data/document: Individual Participant Data Set: SDY625 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY625 — Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort), a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.
- Available data/document: Study Protocol: SDY625 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY625 — ImmPort study identifier is SDY625.
- Available data/document: Study summary, -design, -adverse event(s), -summary of participant assessments, -interventions, -medications, -demographics, -lab tests, -study files, et al.: SDY625 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY625 — ImmPort study identifier is SDY625.